CLINICAL TRIAL: NCT00998556
Title: Effect of Bromocriptine on LV Function in Women With Peripartum Cardiomyopathy A Randomized, Controlled Clinical Trial to Evaluate the Efficacy and Safety of Bromocriptine for Improvement of Left Ventricular Function of Women With PPCM
Brief Title: Effect of Bromocriptine on Left Ventricular Function in Women With Peripartum Cardiomyopathy
Acronym: PPCM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hannover Medical School (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Denise Hilfiker-Kleiner, PhD, Authorized Representative of the Sponsor, Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPCM
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Peripartum Cardiomyopathy
Keywords: Peripartum cardiomyopathy; Bromocriptine
MeSH Terms: conditions — Peripartum Cardiomyopathy | interventions — Bromocriptine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromocriptine (Experimental): Patients randomized to the study medication have to take bromocriptine orally for the first 14 days at a dose of 5 mg/day (= 2 tablets, 1 in morning, 1 in the evening). From day 15 to day 56 they will take a dose of 2.5 mg (= 1 tablet) orally in the evening. The duration of the intervention is 8 weeks, thereafter the patients continue to be observed in the follow-up part of the study up to month 6. The study medication is taken on top of standard therapy for heart failure. Part of this therapy are ACE inhibitors. ACE inhibitors are potentially harmful for the baby when getting into the breast milk, as bromocriptine stops milk production, no additional drug is needed.
  Interventions: Drug: Bromocriptine
- Control Group (No Intervention): The control group will receive standard therapy for heart failure. Part of this therapy are ACE inhibitors. Since ACE inhibitors are potentially harmful for the baby when getting into the breast milk, it is necessary to stop lactation in the control group as well.To stop lactation, application of bromocriptine (2.5mg/day) for up to one week.

INTERVENTIONS:
Drug: Bromocriptine — Patients randomized to the study medication have to take bromocriptine orally for the first 14 days at a dose of 5 mg/day (= 2 tablets, 1 in morning, 1 in the evening). From day 15 to day 56 they will take a dose of 2.5 mg (= 1 tablet) orally in the evening. The duration of the intervention is 8 weeks. The study medication is taken on top of standard therapy for heart failure.
  Arms: Bromocriptine

SUMMARY:
This is a randomized, controlled clinical trial to evaluate the efficacy and safety of bromocriptine for improvement of left ventricular function of women with Peripartum cardiomyopathy (PPCM). A Multi center trial in Germany.

DETAILED DESCRIPTION:
Peripartum cardiomyopathy (PPCM) is a serious life threatening heart disease of unknown etiology in previously healthy women. Only a minority of patients recovers completely while the majority of PPCM patients develop persistent ventricular dysfunction and may experience severe heart failure leading to cardiac transplantation. Thus, these young patients are very sick at a time when the newborn would need a healthy mother. Many of PPCM patients need lifelong treatment causing a large financial and social burden. Indeed, a better understanding of the disease and more efficient therapeutic options are urgently needed. To date, no specific therapy is available so that patients are treated by medical pharmacotherapy for heart failure.

Diagnosis of PPCM is usually made at advanced stages of the disease in severely symptomatic women but prognosis of affected women is poor with reported mortality rates of 15% and recovery in only 23% to 54% of PPCM patients despite optimal medical treatment. Therefore strategies are urgently needed to identify patients at risk and novel therapeutic approaches are required to improve poor prognosis of affected women.

The trial would establish a new specific therapeutic regimen for PPCM and the investigators can expect that such a novel approach would be rapidly adopted in the clinical management of this disease. Since the trial design follows state-of the-art guidelines, the investigators assume that bromocriptine would shortly be adopted into clinical guidelines of the German Cardiac Society, European Cardiac Society, and the American Heart Association.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects in the first 5 months postpartum with new onset of left ventricular (LV) dysfunction (LV ejection fraction ≤35% as assessed by echocardiography) using the internationally accepted criteria for PPCM 1: absence of an identifiable cause of heart failure, absence of recognizable heart disease prior to the last month of pregnancy and LV systolic dysfunction demonstrated by classical echocardiographic criteria.
* Age equal or greater 18
* Written informed consent of the patient

Exclusion Criteria:

* Preexisting cardiac disease (except PPCM which had complete resolution in a previous pregnancy)
* Any preexisting serious conditions
* Previous cardiac surgery or percutaneous coronary intervention
* History of alcohol and/or any other drug abuse
* Contraindication to the planned therapy (e. g. hypersensitivity to trial medication or one of its components)
* Concomitant therapy other than specified in the trial protocol such as products for treatment of fungal infections, psychotropic drugs, medication with the active substances diclofenace, verapamil or doxycycline.
* Women with child bearing potency without effective contraception (i. e. implants, injectables, combined oral contraceptives, some IUDs or vasectomized partner) during the conduct of the trial. Patients using hormonal methods of contraception must be informed about possible influences of the study drug on contraception, in addition heart failure drugs may interfere with contraception. Patients will be counselled about the safest method to be used for contraception.
* Expected low compliance (e.g. by travel distance to trial site)
* Concomitant participation in other clinical trials

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-06; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) from baseline to six months follow-up | 6 months
  Change in left ventricular ejection fraction (LVEF) from baseline to six months follow-up as assessed by cardiac Magnetic Resonance Imaging (MRI) & Echocardiography

SECONDARY OUTCOMES:
Combined endpoint of hospitalization for heart failure, eligibility for cardiac transplantation, cardiac transplantation, and mortality during 6 months follow-up | 6 months
  Combined endpoint of hospitalization for heart failure, eligibility for cardiac transplantation, cardiac transplantation, and mortality during 6 months follow-up; individual components of the combined endpoint; adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Johann Bauersachs, Prof. Dr., Principal Investigator — Hannover Medical School, Hannover, Germany; Denise Hilfiker-Kleiner, Prof. Dr., Study Chair — Hannover Medical School, Hannover, Germany
Locations (1):
- Hannover Medical School (MHH), Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Feyen E, Ricke-Hoch M, Van Fraeyenhove J, Vermeulen Z, Scherr M, Dugaucquier L, Viereck J, Bruyns T, Thum T, Segers VFM, Hilfiker-Kleiner D, De Keulenaer GW. ERBB4 and Multiple MicroRNAs That Target ERBB4 Participate in Pregnancy-Related Cardiomyopathy. Circ Heart Fail. 2021 Jul;14(7):e006898. doi: 10.1161/CIRCHEARTFAILURE.120.006898. Epub 2021 Jul 12. PMID 34247489
- [Derived] Hilfiker-Kleiner D, Haghikia A, Berliner D, Vogel-Claussen J, Schwab J, Franke A, Schwarzkopf M, Ehlermann P, Pfister R, Michels G, Westenfeld R, Stangl V, Kindermann I, Kuhl U, Angermann CE, Schlitt A, Fischer D, Podewski E, Bohm M, Sliwa K, Bauersachs J. Bromocriptine for the treatment of peripartum cardiomyopathy: a multicentre randomized study. Eur Heart J. 2017 Sep 14;38(35):2671-2679. doi: 10.1093/eurheartj/ehx355. PMID 28934837
- [Derived] Haghikia A, Podewski E, Berliner D, Sonnenschein K, Fischer D, Angermann CE, Bohm M, Rontgen P, Bauersachs J, Hilfiker-Kleiner D. Rationale and design of a randomized, controlled multicentre clinical trial to evaluate the effect of bromocriptine on left ventricular function in women with peripartum cardiomyopathy. Clin Res Cardiol. 2015 Nov;104(11):911-7. doi: 10.1007/s00392-015-0869-5. Epub 2015 May 31. PMID 26026286
- See also: If you like to contact us please go to this side and write us an email. We will answer as soon as possible. — http://www.mh-hannover.de/index.php?id=10294&L=1